CLINICAL TRIAL: NCT02997995
Title: A Phase II Trial Testing Durvalumab Combined With Endocrine Therapy in Patients With ER+/Her2- Breast Cancer Eligible for Neoadjuvant Endocrine Therapy And Who Present CD8+ T Cell Infiltration After 4-6 Weeks Exposure to Immune-Attractant
Brief Title: Durvalumab and Endocrine Therapy in ER+/Her2- Breast Cancer After CD8+ Infiltration Effective Immune-Attractant Exposure
Acronym: ULTIMATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Breast International Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0140/1606; UCBG-105 (Other: UNICANCER); BIG 16-01 (Other: BIG); 2016-000764-42 (EudraCT Number)
Record Dates: First submitted 2016-12-09; First posted 2016-12-20 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Estrogen Receptor Positive Tumor; Menopause; Hormone Antagonist
Keywords: T2-T4 Breast cancer; Estrogen Receptor Positive Tumor; PD-1; Neoadjuvant; Immune-attractants; lymphocytes activation
MeSH Terms: conditions — Breast Neoplasms | interventions — tremelimumab; durvalumab; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immune-attractant/lymphocyte activation (Experimental): After the screening phase, the patient will receive immune-attractant combined with exemestane for six weeks. After three weeks (+/- 3 days), a tumor biopsy will be done. Patients who present >10% CD8+ cells in the tumor after 3 weeks and remain eligible will be included in the second part of the trial i.e. lymphocyte activation. In this second part, patients will receive durvalumab 1500 mg Q4W (equivalent to 20 mg/kg Q4W) IV, combined with exemestane (25 mg daily), for six months. The pathological response will be checked by surgery.
  Interventions: Drug: Immune-attractant; Drug: Durvalumab; Procedure: Biopsy

INTERVENTIONS:
Drug: Immune-attractant — The first cohort patients will receive tremelimumab (3 mg/kg, single infusion) as immune-attractants combined with exemestane (25 mg daily).
  Other Names: Tremelimumab
Drug: Durvalumab — Durvalumab (lymphocyte activation) will be administrated at a dose of 1500 mg Q4W (equivalent to 20 mg/kg Q4W) IV, combined with exemestane (25 mg daily), for six months
  Other Names: MEDI4736
Procedure: Biopsy — After three weeks (+/- 3 days) of immune-attractants, a tumor biopsy will be done. Patients who present >10% CD8+ cells in the tumor after 3 weeks will receive the Durvalumab

SUMMARY:
This is an open-label, multicentric, international, phase II trial testing aromatase inhibitors in combination with durvalumab in patients with CD8+ T cell infiltration (>10% CD8+ T cells in the tumor). The trial includes two sequences: The first part of the treatment will consist in 4-6 weeks treatment with immune-attractants; in the second part, CD8+ patients will receive 6 months of durvalumab combined with exemestane.

DETAILED DESCRIPTION:
The study is conducted in 2 parts:

Part 1: lymphocyte attraction. After the screening phase, the patient will receive immune-attractant combined with exemestane for six weeks.

As immune-attractants are added over the course of the study, they will appear as subsequent appendices in the full protocol.

Up to 4 cohorts may be tested sequentially in this design until up to 240 evaluable patients have been treated.

The first cohort of patients will receive tremelimumab (3 mg/kg, single infusion) combined with exemestane (25 mg daily). In each cohort, an interim analysis will be performed after 30 patients in order to potentially stop the cohort (if less than 25% of patients present >10% CD8+ cells in the tumor after 3 weeks). If all 4 cohorts are closed and the target number of 56 patients for part 2 has not been reached, additional patients will be recruited and treated with the best performing immune-attractant treatment based on the part I results. From the moment 56 patients are included in part 2, no more patients will be entered in part 1.

After three weeks (+/- 3 days), a tumor biopsy will be done. Patients who present >10% CD8+ cells in the tumor after 3 weeks and remain eligible will be included in the second part of the trial (patients who do not present CD8+ T cells on the 3-week biopsy will be treated at the investigator's choice).

Part 2: lymphocyte activation (anti-PD1 treatment) Four to six weeks after immune-attractant start, patients having >10% CD8+ cells in the tumor will receive durvalumab 1500 mg Q4W (equivalent to 20 mg/kg Q4W) IV, combined with exemestane (25 mg daily), for six months.

Part 2 will include two steps. In the first step, we will include 23 patients. If 2 or more pathological complete responses are observed in these 23 patients, the part 2 will move to step 2. 33 additional patients will be included in the step 2.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years post-menopausal according to one of the following criteria:

   * Age >60 years
   * Or Bilateral ovariectomy
   * Or Age ≤60, with an uterus and presenting an amenorrhea of more than 12 months and FSH and estradiol in the postmenopausal range
   * Or Age ≤60, without an uterus and FSH and estradiol in the postmenopausal range
2. Histologically proven invasive breast cancer eligible to neoadjuvant endocrine therapy according to multidisciplinary tumor board.

   Note: Multicentric/multifocal tumors are allowed if all share the same characteristics
3. cT2-T4, any N; cT2 are eligible only if the clinical tumor size is >3 cm
4. Non metastatic, M0 (according to clinical staging)
5. Luminal A patients ER-positive by immunohistochemistry (IHC) according to the following criteria (local assessment): Grade I or II AND ER-positive (≥60%) AND Ki67 <20%
6. Her2-negative by IHC (score 0 or 1+) and/or fluorescent in situ hybridization (FISH)/chromogenic in situ hybridization (CISH) negative according to local assessment
7. CD8+ T Cell infiltration defined as >10% cells stained with anti-CD8 monoclonal antibody by IHC at the 3-week biopsy (applicable for inclusion in part 2 only)
8. Available tumor samples from baseline biopsy
9. World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrolment
10. Adequate organ and marrow function as defined below:

    * Hemoglobin ≥9.0 g/dL
    * Absolute neutrophil count ≥1.5 × 10⁹/L
    * Platelet count ≥100 × 10⁹/L
    * Serum bilirubin ≤1.5 × upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome, who will be allowed in consultation with their physician
    * Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤2.5 × ULN
    * Adequate renal function as determined by CKD-EPI formula (using actual body weight)
11. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures
12. Written informed consent obtained prior to performing any protocol-related procedures, including screening evaluations

Exclusion Criteria:

1. Inflammatory breast cancer
2. No prior exposure to immune-mediated therapy including, but not limited to, other anti-CTLA-4, anti-PD-1, anti-PD-L1, and anti-programmed cell death ligand 2 (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines
3. Any concurrent chemotherapy, investigational product (IP), biologic therapy for cancer treatment
4. Previous Radiotherapy treatment to more than 30% of the bone marrow;
5. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose
6. History of allogenic organ transplantation
7. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis with the exception of diverticulosis, celiac disease or other serious gastrointestinal chronic conditions associated with diarrhea), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis), Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement or psoriasis not requiring systemic treatment
8. Any condition that, in the opinion of the Investigator, would interfere with the evaluation of investigational product or interpretation of patient safety or study results, including ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events from investigational products, or compromise the ability of the patient to give written informed consent
9. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms
10. History of active primary immunodeficiency
11. Known history of active tuberculosis
12. Active infection including hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
13. Current or prior use of immunosuppressive medication within 14 days before the first dose. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection)
    * Systemic corticosteroids at physiologic doses not exceeding 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
14. Receipt of live, attenuated vaccine within 30 days prior to the first dose of IP.

    Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of IP
15. Known allergy or hypersensitivity to any medicinal product used in the trial or any excipient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
pathological Complete Response | at time of surgery
  Response at surgery

SECONDARY OUTCOMES:
Number of CD8+ T cell | at biopsy (3 weeks)
  exam at biopsy and comparison between biopsy and Baseline biopsy rates
Clinical response | after 6 months of Durvalumab
  Clinical exam
Assessment of Ki67 | at surgery
  measure of Ki67
Toxicities | 1 year and 8 months
  Common terminology criteria for adverse events (CTC-AE) v4.03
Predictive value of Mutational load for efficacy of Durvalumab | on baseline biopsy and blood samples
  exome sequencing on baseline samples
Predictive value of PDL1 expression for the efficacy of Durvalumab | on baseline biopsy and biopsy at 3 weeks
  correlate Immune infiltrate intensity with the proportion of tumor cells expressing PD-L1 by Ventana SP263 assay

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Andre, Prof, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (29):
- France (21):
  - Centre Hospitalier cote Basque, Bayonne
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Hospitalier de Cahors, Cahors
  - Centre Hôspitalier de Cholet, Cholet
  - Centre George François Leclerc, Dijon
  - Institut Daniel Hollard Groupe Hôspitalier, Grenoble
  - Centre Oscar Lambret, Lille
  - CHU Limoges, Limoges
  - Centre Hospitalier Bretagne Sud, Lorient
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut Curie Site Paris, Paris
  - Hôpital Saint Louis APHP, Paris
  - Centre Hospitalier Perpignan, Perpignan
  - Institut Jean Godinot, Reims
  - Institut Curie Hôpital René Huguenin, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - CHU Bretonneau - Centre Henry Kaplan, Tours
  - Gustave Roussy, Villejuif
- Spain (7):
  - ICO Badalona, Badalona
  - Hospital Clinic Barcelona, Barcelona
  - HU Vall Hebron, Barcelona
  - HU Arnau de Vilanova, Lleida
  - CIO Clara Campal, Madrid
  - HU Ramon y Cajal, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided